CLINICAL TRIAL: NCT01094067
Title: Multi-center, Double-blind, Randomized, Placebo-controlled, Cross-over Study to Demonstrate That a Single Infusion of Tezosentan Has Minimal Effect on Blood Pressure in Patients With Pulmonary Arterial Hypertension, Treated With Endothelin Receptor Antagonists, Phosphodiesterase-5 Inhibitors or a Combination of Both.
Brief Title: Tezosentan in Patients With Pulmonary Arterial Hypertension
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow recruitment, the study was prematurely discontinued.
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: AC-051-207
Record Dates: First submitted 2010-03-25; First posted 2010-03-26 (Estimated); Last update posted 2018-07-09 (Actual); Status verified 2018-07

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Placebo at visit 1, tezosentan at visit 2
  Interventions: Drug: ACT-050089; Other: Placebo
- 2 (Experimental): Tezosentan at visit 1, placebo at visit 2
  Interventions: Drug: ACT-050089; Other: Placebo

INTERVENTIONS:
Drug: ACT-050089 — 5 mg/h intravenously, Tezosentan
Other: Placebo — Matching placebo

SUMMARY:
Multicenter, double-blind, randomized, placebo-controlled, cross-over study to demonstrate that a single infusion of tezosentan has minimal effect on blood pressure in patients with pulmonary arterial hypertension, treated with endothelin receptor antagonists, phosphodiesterase-5 inhibitors or a combination of both.

ELIGIBILITY:
Inclusion Criteria :

1. Signed informed consent prior to initiation of any study-mandated procedure
2. Male and female patients 18 years of age or older
3. Patients with PAH according to one of the following subgroups of the Dana Point Classification Group 1:

   * Idiopathic, or
   * Heritable, or
   * Associated with connective tissue disease
4. Documented hemodynamic diagnosis of PAH by right heart catheterization (not part of study mandated procedures):

   * Resting mean pulmonary arterial pressure (mPAP) ≥ 25 mmHg and
   * Resting mean pulmonary vascular resistance (PVR) ≥ 240 dyn•s•cm 5 and
   * Pulmonary capillary wedge pressure ≤ 15 mmHg
5. Modified NYHA functional class II-III
6. Patients on treatment with ERAs, PDE-5 inhibitors or a combination of both, if used for at least 3 months prior to Visit 1 and dosing kept stable for at least 28 days prior to Visit 1.

Exclusion Criteria :

1. Patients with PAH in Dana Point Classification Groups 2-5, and PAH Group 1 subgroups not covered by inclusion criterion No. 3
2. Patients with sitting SBP < 100 mmHg
3. Patients with sitting DBP < 60 mmHg
4. Patients with body weight < 50 kg (110 lbs)
5. Patients with clinically significantly elevated liver enzymes (AST, ALT and/or alkaline phosphatase > 3 times upper limit)
6. Patients with clinically significant chronic renal insufficiency (serum creatinine >2.5mg/dL / 221 µmol/L)
7. Patients with moderate or severe hepatic impairment (Child-Pugh B and C)
8. Patients who have received prostacyclin (epoprostenol) or prostacyclin analogs (e.g., treprostinil, iloprost and beraprost) within 28 days of Visit 1
9. Patients who have received any investigational drugs within 28 days of Visit 1
10. Patients who have received cyclosporine A (CsA) or tacrolimus within 28 days of Visit 1
11. Psychotic, addictive or other disorder limiting the ability to provide informed consent or to comply with the study
12. Life expectancy less than 12 months
13. Females who are lactating or pregnant (positive pre-treatment pregnancy tests) (serum test at Screening and urine test on Visit 1 and 2) or females who are not using a reliable method of birth control (failure rate less than 1% per year) during the study and for at least one month after last administration of study drug
14. Known hypersensitivity to any of the excipients of the drug formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2010-09-01; Primary Completion 2010-12-01 (Actual); Study Completion 2011-09-01 (Actual)

PRIMARY OUTCOMES:
Absolute change in supine SBP from Baseline to 30 minutes at each visit (Visit 1 and Visit 2) - in mmHg | 30 days

SECONDARY OUTCOMES:
Absolute change in heart rate from Baseline to 30 minutes at each visit (Visit 1 and Visit 2) - in bpm | 30 days

CONTACTS AND LOCATIONS:
Locations (5):
- Baylor College of Medicine, Houston, Texas, United States
- Hopital Antoine Beclere, Clamart, France
- Japan (3):
  - Osaka University Hospital, Osaka
  - National Cardiovascular Center, Osaka
  - Keio University Hospital, Shinjuku-Ku